CLINICAL TRIAL: NCT05117398
Title: Randomized Open-label Controlled Trial Evaluating a Single-dose Intravenous Dalbavancin Versus Standard Antibiotic Therapy During Catheter-related Bloodstream Infections Due to Staphylococcus Aureus
Brief Title: Dalbavancin Versus Standard Antibiotic Therapy for Catheter-related Bloodstream Infections Due to Staphylococcus Aureus
Acronym: DALICATH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre Hospitalier de Perigueux (Other); Advanz Pharma (Industry); Nantes University Hospital (Other); Centre National de Référence des staphylocoques (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220763; 2021-004038-12 (EudraCT Number)
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Catheter Bacteremia; Staphylococcus Aureus Infection
Keywords: catheter-related bloodstream infections; Staphylococcus aureus infection
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: Phase III, pragmatic, open-label, non-inferiority, randomized (1:1), multicenter trial, in patients with non-complicated CR-BSI due to S. aureus, with two parallel groups receiving 14 days of active antimicrobial therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dalbavancin (Experimental): Dalbavancin (Xydalba®) 1500 mg - One unique dose
  Interventions: Drug: Dalbavancin administration
- Standard documented antibiotic therapy for 14 days according to national guidelines. (Active Comparator): As currently recommended, investigators will be encouraged to use the intravenous route for the entire duration of treatment. However, in order to interfere as little as possible with usual practice in each center, the antimicrobial therapy will be let to the choice of the physician in charge of the patient after a minimum of 7 days of intravenous treatment.
  During all the duration of the study, in case of worsening of the clinical condition requiring the prescription of antistaphylococcal, the clinician will prescribe additional antibiotherapy according to standard good practice.
  Interventions: Drug: Standard antibiotic therapy

INTERVENTIONS:
Drug: Dalbavancin administration — A single-dose of intraveneuse (IV) administration of dalbavancin of 1500 mg.
  In case of patients with chronic renal impairment (creatinin clairance < 30mL/min), a single-dose of IV administration of reduced dalbavancin of 1000 mg.
  Other Names: Xydalba® administration
  Arms: Dalbavancin
Drug: Standard antibiotic therapy — Standard Antibiotic therapy according to national recommendations. During the study, the start of treatment is considered to be the day of inclusion/randomization (even if active antiobiotic treatment was started, less than 72 hours ago according to inclusion criteria).
  Other Names: Standard documented antibiotic therapy
  Arms: Standard documented antibiotic therapy for 14 days according to national guidelines.

SUMMARY:
The primary objective of the study is to demonstrate, among patients with non-complicated CR-BSIs due to S. aureus, that a single-dose of intravenous (IV) dalbavancin 1500 mg is non-inferior to standard documented antibiotic therapy for 14 days according to national guidelines at DAY 30 (Long follow up visit).

As the secondary objectives, the study aims to evaluate according to treatment group:

1. Cure rate at DAY 14 and DAY 90 (EOS);
2. Mortality rate within 90 days of follow-up;
3. Time to negativation of blood cultures;
4. Patient's quality of life;
5. Hospitalization length of stay;
6. Cost-utility analyses;
7. Occurrence of any adverse event (AE and SAE), until Day 90 (EOS).

DETAILED DESCRIPTION:
Catheter-related bloodstream infections (CR-BSIs) are the most common nosocomial bloodstream infections, with an incidence as high as 8.5 to 19.8 infections per 1000 catheter-days. Staphylococcus aureus is involved in about 20% of CR-BSIs and associated with significant morbidity, mortality (9.3%), prolonged hospital stay (+ 9 days), and healthcare costs (35 000 € to 65 000 € per case). S. aureus CR-BSIs occurs mainly in frail patients with a port of catheter for chemotherapy or parenteral nutrition.

According to international guidelines, management of CR-BSIs due to S. aureus includes the removal and replacement of the infected catheter and a 14-day intravenous (IV) antibiotic therapy. Therefore, the management of CR-BSIs due to S. aureus requires the insertion of a new intravenous catheter. In turn, the new catheter can also lead to new septic complications and limit the patients' autonomy. Non-adherence to these recommendations leads to over-mortality and costs.

Following of the positive results of the SABATO trial in 2021 to determine whether early switch to oral antibiotic therapy is safe and effective in patients with uncomplicated BSA, oral switch during staphylococcal bacteremia, will likely become the standard of care. It is therefore justified to allow oral switch in the control arm.

The usual practice in some centers is already to switch to oral antibiotics, after a minimum of 7 days of intravenous treatment.

Dalbavancin is a new glycopeptide antibiotic, with an excellent bactericidal activity against Gram-positive bacteria, especially S. aureus, and a prolonged half-life of 14 to 15 days. As a comparison, half-life of antibiotics usually used for CR-BSIs due to S. aureus, i.e. penicillin or glycopeptide, as-per sensitivity to methicillin is much lower: 1.5 to 9 hours. Such prolonged half-life allows one IV injection to be sufficient and effective over 14 days of treatment. This remarkable characteristic should allow patients to be promptly discharged from hospital without monitoring.

The hypothesis of the study is that in patients with CR-BSIs due to S. aureus, after catheter removal, dalbavancin could be administered intravenously in a single administration after catheter removal and be as effective as standard documented antibiotic therapy for 14 days according to national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years;
* Blood cultures positive for S. aureus, obtained within 72 hours before randomization (the date considered is the date of the sampling, not the results);
* CR-BSI, defined as:

  * One positive blood culture AND Local signs of infection at the catheter site; OR
  * at least one positive blood culture obtained from the catheter and the peripheral vein; AND
  * A differential period between catheter versus peripheral blood culture positivity of at least 2h as recommended; AND
  * Same S. aureus isolate (same phenotype) identified from the catheter and the peripheral vein blood cultures; OR
  * One positive blood culture; AND
  * Strong presumption of catheter-related infection according to clinical opinion.
* Intravascular catheter - implantable venous access device (port-a-cath and Piccline) - removed before randomization;
* Informed consent form date and signed by the patient.

Exclusion Criteria:

* Polymicrobial infection;
* Dalbavancin resistant strain;
* More than 72 hours of active antibiotic treatment targeting S. aureus (in-vitro susceptibility) administered prior to randomization;
* Patient with known valvulopathy, previous history of endocarditis, or suspicion of infective endocarditis by physician in charge;
* Suspicion of any other deep focus infections, such as arthritis, pneumonia, osteomyelitis, or meningitis, presence of cerebral or peripheral emboli (arterial occlusion);
* Thrombophlebitis;
* Failure to remove any intravascular catheter which was present when first positive blood culture;
* Signs of infection associated with quick SOFA score ≥ 2 at randomization;
* Patients with foreign bodies such as: prosthetic heart valve, endovascular prosthesis, ventriculo-atrial shunt, pacemaker, or an automated implantable cardioverter defibrillator (AICD) device;
* Severe liver disease (Child-Pugh C);
* Severely immunocompromised patients:

  * Neutropenia (< 500 neutrophils/µL) at randomization;
  * Hematopoietic stem cell transplantation within the past 6 months or planned during treatment period;
  * Solid organ transplant;
* Contraindication to dalbavancin and/or glycopeptide;
* Life expectancy < 3 months;
* Active injection drug user;
* Pregnant or breastfeeding women;
* For premenopausal women: failure to use highly-effective contraceptive methods for 1 month after receiving study drug;
* Participation in other interventional trials ongoing;
* Persons held in an institution by legal or official order;
* Patients under legal protection;
* Patients under guardianship or curators;
* Patients unable to give a free and informed consent;
* Patient not affiliated to a social security scheme: obligation of affiliation to a social security scheme or to be a beneficiary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Cure rate | DAY 30
  Clinical cure without relapse, defined by the absence of all the following:
  * Local and/or general signs of infection:
  * Relapse of bacteremia to S. aureus - i.e. a bacteremia due to S. aureus occurring after initial negativation of blood cultures (2 vials);
  * In dalbavancin arm: Any additional antibiotic therapy active on S. aureus received between DAY 0 and DAY 14;
  * In both arms: Any additional antibiotic therapy active on S. aureus received after DAY 14; i.e. between DAY 14 and DAY 30;
  * Deep focus infection including endocarditis;
  * Death from all causes.

SECONDARY OUTCOMES:
Cure rate | DAY 14;DAY 90 (EOS)
  Clinical cure at DAY 14 and DAY 90 (EOS) defined by the absence of all the following:
  * For DAY 14 and DAY 90:
    a. Local and/or general signs of infection: i. local: redness, induration, swelling, purulent discharge; ii. general: fever, chills; b. Relapse of bacteremia to S. aureus - i.e. a bacteremia due to S. aureus occurring after initial negativation of blood cultures (2 vials);
  * Additional criteria at EOS only:
    c. Any additional antibiotic therapy active on S. aureus received between DAY 14 and DAY 90 (EOS);
Mortality rate | DAY 90
  Death all-cause occurring within 90 days of follow-up.
Bloodstream clearance | DAY 14
  Time from first positive blood culture to first negative blood cultures (in days), limited to DAY 14.
Patient's quality of life | BASELINE; DAY 14; DAY 30; DAY 90 (EOS)
  Autonomy, pain and anxiety using 5-level EQ-5D scale
Hospitalization length of stay | DAY 90
  Hospitalization duration in days
Cost-utility analyses | DAY 90
  Cost per avoided relapse; life-year gained, and per quality-adjusted life year (QALY)
Incidence of any adverse event (AE and SAE) | DAY 90
  Proportion of patients with any adverse event until the end of study. It includes the complications due to venous catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard CASTAN, MD, Principal Investigator — CH de Perigueux; Aurélien DINH, MD, PhD, Study Director — APHP - RAYMOND POINCARE
Locations (2):
- France (2):
  - Infectious Diseases Department, Raymond-Poincaré Hospital - APHP, Garches
  - Infectious Diseases Department, CH PERIGUEUX, Périgueux

IPD SHARING:
Plan to Share IPD: No